CLINICAL TRIAL: NCT02661945
Title: Usefulness of Near-focus With Narrow-band Imaging for Determining Gastric Tumor Margin
Brief Title: Usefulness of Near-focus With Narrow-band Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Wook Kim, Assistant Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NFNBI
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Gastric Tumors
Keywords: near focus with narrow band imaging; tumor margin; indigocarmine chromoendoscopy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Narrow Band Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Near focus with narrow band imaging (Experimental): Near focus with narrow band imaging is used for marking the tumor margin.
  Interventions: Device: Near focus with narrow band imaging
- Indigo carmin (No Intervention): After indigo carmine was sprayed over the lesion, marking is performed.

INTERVENTIONS:
Device: Near focus with narrow band imaging
  Arms: Near focus with narrow band imaging

SUMMARY:
Near-focus with narrow-band imaging is a novel technique to improve the quality of images of the irregular mucosal structures and microvessels of gastric neoplasms. The investigators compare this technique with indio carmin spray, commonly used tool to determine tumor margin. The subject are patients who underwent endoscopic submucosal dissection for gastric neoplasms. Participants are randomized into near-focus with narrow-band imaging and indigo carmin groups. First, marking is performed at the tumor margins determined by each modality. The distance from the marking dots to the tumor margin is measured histopathologically in the resected specimens. Finally, the investigators will compare the accuracy between two groups based on the distance from marking dots to tumor margin measured by histopathologic examination.

ELIGIBILITY:
Inclusion Criteria:

* Participants who undergo endoscopic submucosal dissection for gastric tumors (early gastric carcinoma or gastric adenoma)

Exclusion Criteria:

* fail to en bloc resection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Accuracy (accurate if the distance (between margin dots and tumor margin measured by histopathology) was less than 1 mm) | 1 week after procedure
  Marking was diagnosed as accurate if the distance (between margin dots and tumor margin measured by histopathology) was less than 1 mm

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Cheonan Hospital, Soonchunhyang University College of Medicine, Cheonan, Chungcheongnam-do
  - Korea University Medical Center, Seoul, Seongbuk-gu
  - Inha University School of Medicine, Incheon
  - Pusan National University School of Medicine, Pusan
  - Kyung Hee University Hospital, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Seoul
  - Soonchunhyang University Hospital, Seoul

REFERENCES:
- [Background] Nagahama T, Yao K, Maki S, Yasaka M, Takaki Y, Matsui T, Tanabe H, Iwashita A, Ota A. Usefulness of magnifying endoscopy with narrow-band imaging for determining the horizontal extent of early gastric cancer when there is an unclear margin by chromoendoscopy (with video). Gastrointest Endosc. 2011 Dec;74(6):1259-67. doi: 10.1016/j.gie.2011.09.005. PMID 22136775
- [Result] Kiyotoki S, Nishikawa J, Satake M, Fukagawa Y, Shirai Y, Hamabe K, Saito M, Okamoto T, Sakaida I. Usefulness of magnifying endoscopy with narrow-band imaging for determining gastric tumor margin. J Gastroenterol Hepatol. 2010 Oct;25(10):1636-41. doi: 10.1111/j.1440-1746.2010.06379.x. PMID 20880172
- [Derived] Kim JW, Jung Y, Jang JY, Kim GH, Bang BW, Park JC, Choi HS, Cho JH; Research Group for Endoscopic Instruments and Stents of Korean Society of Gastrointestinal Endoscopy. Narrowband imaging with near-focus magnification for discriminating the gastric tumor margin before endoscopic resection: A prospective randomized multicenter trial. J Gastroenterol Hepatol. 2020 Nov;35(11):1930-1937. doi: 10.1111/jgh.15109. Epub 2020 Jun 16. PMID 32433790